CLINICAL TRIAL: NCT04585191
Title: Reducing Treatment Risk in Older Patients With Diabetes: Comparative Effectiveness of Academic Detailing With and Without Pre-Visit Patient Preparation
Brief Title: Reducing Treatment Risk in Older Adults With Diabetes
Acronym: RETRO-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CDR-2019C1-16126
Record Dates: First submitted 2020-09-28; First posted 2020-10-14 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes Treated With Insulin; Hypoglycemia; Primary Health Care; Polypharmacy
Keywords: clinical trial
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Intervention Model Description: There are two arms within the Comparative Effectiveness Randomized Clinical Trial (CE-RCT). All eligible primary care physicians (PCPs) will receive academic detailing. Eligible and consenting patients of these PCPs will be randomly allocated to intervention vs attention control arms grouped by PCP. (There will be a secondary, parallel comparison group to measure temporal trends in care for similar patients at other facilities in our care system not involved in the clinical trial.)
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Visit Conversation Aid (Experimental): Patients in the intervention arm will receive a newly developed, 1-page conversation aid/communication tool entitled "Talking to Your Doctor about Diabetes: Are My Current Medicines Still Right for Me?" prior to a scheduled appointment with their primary care physician (PCP). This document will provide brief education about changing risks and benefits of diabetes treatment as patients age, elicit values and preferences regarding treatment, and help direct next conversation steps.
  Interventions: Behavioral: Conversation Aid
- General Health Education Handout (Active Comparator): Patients in the attention control arm will receive an existing 1-page health education handout entitled "Embracing Life as You Age" which provides some general advice geared towards older patients such as remaining physically active, limiting sun exposure, and eating well.
  Interventions: Other: Attention Control Educational Handout

INTERVENTIONS:
Behavioral: Conversation Aid — Intervention is a newly developed, 1-page conversation aid/communication tool entitled "Talking to Your Doctor about Diabetes: Are My Current Medicines Still Right for Me?" that patients receive prior to a scheduled appointment with their primary care physician (PCP). This document will provide brief education about changing risks and benefits of diabetes treatment as patients age, elicit values and preferences regarding treatment, and help direct next conversation steps.
  Arms: Pre-Visit Conversation Aid
Other: Attention Control Educational Handout — Attention control is an existing health education handout that provides some general health advice geared towards older patients.
  Arms: General Health Education Handout

SUMMARY:
This study will evaluate the impact of academic detailing (evidence-based provider education) with or without patient pre-visit preparation (elicitation of values and preferences) on safe insulin de-prescribing among older patients with type 2 diabetes at risk for hypoglycemia. The hypothesis is that patients who are well-prepared for their primary care visit will engage in more informed discussions with their providers regarding re-evaluation of current treatment regimens. In clinically appropriate cases, these more effective discussions will result in safe de-prescribing and fewer future episodes of hypoglycemia.

DETAILED DESCRIPTION:
In this comparative effectiveness clinical trial, primary care physicians (PCPs) will receive 2 academic detailing sessions 6 months apart. Eligible patients (age 75 years or greater, type 2 diabetes, prescribed insulin or sulfonylureas [SUs], and last measured HbA1c <=8%) of these PCPs will be randomized to receive either a pre-visit conversation aid/communication tool that elicits values and preferences regarding safe insulin/SU deprescribing [Intervention] or a general health education handout ("Embracing Life as You Age") [Attention Control]. Patient-reported outcomes (e.g., self-reported hypoglycemia episodes) and clinical outcomes (e.g., changes in glycemic regimen) will be compared between study arms. If successful, this study will provide evidence to support strategies for safer treatment in older adults with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 75 years
* type 2 diabetes with last measured Hemoglobin A1c (HbA1c) ≤ 8.0%
* currently prescribed insulin and/or sulfonylureas (SUs)
* Kaiser Permanente Northern California member

Exclusion Criteria:

* Given the requirements of this funding mechanism, we will not be able to develop new patient materials in languages other than English, and patients unable to communicate in English will be excluded.
* Similarly, patients unable to provide informed consent and/or participate in informed decision making due to cognitive or communication-related deficits will be excluded.
* Excluded by their primary care provider

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 450 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Grant, MD MPH, Principal Investigator — Division of Research, Kaiser Permanente Northern California
Locations (4):
- United States (4):
  - Kaiser Permanente South San Francisco, San Francisco, California
  - Kaiser Permanente Northern California, San Leandro, California
  - Kaiser Permanente Union City, Union City, California
  - Kaiser Permanente Vallejo, Vallejo, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grant RW, Peterson I, McCloskey JM, Lipska KJ, Nugent J, Karter AJ, Gilliam LK. Diabetes Deprescribing in Older Adults: A Randomized Clinical Trial. JAMA Intern Med. 2025 Aug 1;185(8):926-935. doi: 10.1001/jamainternmed.2025.2015. PMID 40549370

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients provided informed consent and were enrolled into the study. All study outcomes are measured at the patient level, with clustering within primary care physician panel accounted for in all outcome analyses.
Pre-assignment Details: Among primary care physicians (PCPs) who attended the academic detailing sessions, their study eligible patients provided informed consent, were enrolled in the study, and are the subject of all outcome analyses. PCPs assented to participate but were not asked to provide informed consent and are therefore not considered the primary subjects of this RCT.
Groups:
- Pre-Visit Conversation Aid: Patients in the intervention arm will receive a newly developed, 1-page conversation aid/communication tool entitled "Talking to Your Doctor about Diabetes: Are My Current Medicines Still Right for Me?" prior to a scheduled appointment with their PCP. This document will provide brief education about changing risks and benefits of diabetes treatment as patients age, elicit values and preferences regarding treatment, and help direct next conversation steps.
  Conversation Aid: Intervention is a newly developed, 1-page conversation aid/communication tool entitled "Talking to Your Doctor about Diabetes: Are My Current Medicines Still Right for Me?" that patients receive prior to a scheduled appointment with their PCP. This document will provide brief education about changing risks and benefits of diabetes treatment as patients age, elicit values and preferences regarding treatment, and help direct next conversation steps.
Period: Overall Study
Arm/Group | Pre-Visit Conversation Aid | General Health Education Handout
Started | 232 | 218
Completed | 232 | 218
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-Visit Conversation Aid | General Health Education Handout | Total
Number analyzed (Participants) | 232 | 218 | 450
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 232 | 218 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.7 (3.9) | 80.2 (4.2) | 79.9 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 112 | 223
  Male | 121 | 106 | 227
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 35 | 42 | 77
  Black/African-American | 32 | 29 | 61
  Asian | 39 | 34 | 73
  Multi/Other | 15 | 11 | 26
  Missing/Unknown | 1 | 1 | 2
  White | 110 | 101 | 211
Region of Enrollment [Number; unit: participants]
  United States | 232 | 218 | 450

OUTCOME MEASURES:

1. Primary Outcome: Clinical Outcome: Number of Participants With Glycemic Regimen De-prescribing
Description: Aggregate binary measure of diabetes medication deprescribing between baseline and 6-month follow-up. Greater de-prescribing is better.
  De-prescribing defined as any combination of:
  1. Discontinuation of either insulin or a sulfonylureas (SU)
  2. Reduction in dose of insulin or SU,
  3. Switch from a higher risk to lower risk version of insulin (e.g. from sliding scale insulin or basal-bolus insulin to twice daily basal insulin) and/or higher risk to lower risk oral medicine (e.g. switching from SU to other oral medicine less associated with hypoglycemia).
Time Frame: 6 months after initial primary care visit
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Visit Conversation Aid | General Health Education Handout
Number analyzed (Participants) | 232 | 218
Participants | 34 | 21

2. Primary Outcome: Patient-Reported Outcome: Number of Participants With Self-Reported Hypoglycemia
Description: Patient report of any low blood sugar episode in past 6 months that resulted in passing out or needing help from someone else
Time Frame: Preceding 6 month period (asked 6 months after initial primary care visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Visit Conversation Aid | General Health Education Handout
Number analyzed (Participants) | 232 | 218
Participants | 10 | 13

3. Secondary Outcome: Diabetes Treatment Satisfaction Questionnaire Scores
Description: Patient-Centered Outcome: Number of Participants with improved scores on Diabetes Treatment Satisfaction Questionnaire [8 items, scores 0 - 36, higher score is better]
Time Frame: Asked 6 months after initial primary care visit
Reporting Status: Not Posted, anticipated posting 2025-05

4. Secondary Outcome: Number of Participants With Hypoglycemic-related Hospitalizations
Description: Hypoglycemic-related hospitalizations in the 6 months following the first study-related visit.
Time Frame: 6 months following the first study-related visit
Reporting Status: Not Posted

5. Secondary Outcome: RAND Patient Satisfaction Questionnaire
Description: Patient-Centered Outcome: Number of Participants with improved scores on the RAND Patient Satisfaction Questionnaire [5 item, score 5- 25, higher is worse]
Time Frame: 6 months following the first study-related visit
Reporting Status: Not Posted, anticipated posting 2025-05

6. Secondary Outcome: Perceived Efficacy in Patient - Physician Interactions
Description: Patient-Centered Outcome: Number of Participants with improved scores on Perceived Efficacy in Patient - Physician Interactions (5 - Item Survey, score 5-25, higher is better)
Time Frame: 6 months following the first study-related visit
Reporting Status: Not Posted, anticipated posting 2025-05

7. Other Pre Specified Outcome: Change in HbA1c Level
Description: HbA1c Change from baseline to study completion, an average of 1 year
Time Frame: 1 year following the first study-related visit
Reporting Status: Not Posted, anticipated posting 2025-05

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Pre-Visit Conversation Aid | General Health Education Handout
All-Cause Mortality (participants affected / at risk) | 7/232 | 10/218
Serious Adverse Events (participants affected / at risk) | 0/232 | 0/218
Other Adverse Events (participants affected / at risk) | 0/232 | 0/218

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT04585191/Prot_SAP_000.pdf